CLINICAL TRIAL: NCT07133087
Title: Body Awareness, Upper Extremity Function, and Quality of Life in Breast Cancer Survivors: A Case-Control Study
Brief Title: Body Awareness, Upper Extremity Function, and Quality of Life in Breast Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Other Study IDs: ssaka10
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; body awareness
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control group: A group of healthy subjects, matched with the breast cancer group based on criteria such as age and body mass index, will be included in the study.
- Breast cancer group: Women who have survived Stage 0-III breast cancer will be included in the study.

SUMMARY:
Breast cancer is one of the most common types of cancer among women and one of the leading causes of morbidity and mortality. With increasing survival rates, issues such as treatment-related morbidities and consequently upper extremity dysfunction, reduced body awareness, and decreased quality of life are frequently encountered. In the literature, the impact of treatment-related morbidities-particularly on upper extremity functions, body awareness, and quality of life-among women who have survived breast cancer treatment has not been sufficiently investigated. This gap constitutes a significant shortcoming in terms of clinical practices and the post-treatment period.

This study aims to examine the effects of breast cancer treatment on upper extremity functions, body awareness, and quality of life in women who have survived breast cancer treatment, in comparison with a healthy control group. The study will be conducted at Yeditepe University Koşuyolu Hospital between May, 2025, and October, 2025. Participants will include women who have survived breast cancer treatment and a healthy control group matched based on criteria such as age and body mass index.

In the study, three separate assessments will be conducted for upper extremity functions: the "Quick Disabilities of the Arm, Shoulder, and Hand" (QuickDASH) questionnaire for upper extremity functionality, a hand dynamometer for grip strength, and the Clinometer device for shoulder joint position sense. The "Body Awareness Questionnaire" will be used to assess body awareness, and the "EORTC QLQ-C30" scale will be used for quality of life assessment. The IBM SPSS Statistics software package will be used for data analysis. In statistical analyses, a significance level of p<0.05 will be considered.

ELIGIBILITY:
Inclusion Criteria for breast cancer survivors:

* Being a woman
* Being between the ages of 25 and 75
* Having been diagnosed with Stage 0-III breast cancer
* Having completed primary treatments (surgery, chemotherapy, and/or radiation therapy) no more than 6 months prior to the assessment date
* Having received medical clearance from a physician
* Having undergone either breast-conserving surgery or mastectomy due to breast cancer
* Willingness to participate in the study voluntarily

Exclusion Criteria for breast cancer survivors:

* Having a history of rehabilitation due to upper extremity, thoracic, or cervical musculoskeletal disorders within 6 months prior to the breast cancer diagnosis
* Having a history of neuromuscular dysfunction
* Using medications that may affect neuromuscular performance

Inclusion criteria for the control group:

* Being a woman
* Having a body mass index (BMI) within ±3 kg/m² of the breast cancer survivor group
* Being within ±5 years of age compared to the breast cancer survivor group
* Matching hand dominance with the breast cancer survivor group

Exclusion criteria for the control group:

* Having a history of neuromuscular dysfunction
* Using medications that may affect neuromuscular performance
* Having a history of rehabilitation due to upper extremity, thoracic, or cervical musculoskeletal disorders within the last 6 months

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of women who have survived breast cancer treatment at Yeditepe University Koşuyolu Hospital and a healthy control group. The sample will include breast cancer survivors and healthy controls who meet the inclusion and exclusion criteria and voluntarily agree to participate in the study.
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Body Awareness Scale | At the day of enrollment
  The scale consists of 18 items evaluated on a 7-point Likert scale and aims to determine the sensitivity level of body composition through 4 subgroups. The four sub-parameters of the scale are: "Changes in Body Processes," "Sleep-Wake Cycle," "Prediction of Illness Onset," and "Prediction of Bodily Reactions."
Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire | At the day of enrollment
  The questionnaire will be used to determine individuals' levels of functionality.
Hand Grip Strength Assessment | At the day of enrollment
  A Jamar Hand Dynamometer (Takei Scientific Instruments Co., Ltd - Japan) will be used to measure participants' maximum grip strength
Shoulder Joint Position Sense | At the day of enrollment
  Shoulder joint position sense will be assessed using the "Clinometer" smartphone application. Goniometer and inclinometer applications, adapted for both iOS and Android systems, are low-cost methods with proven validity and reliability, accessible to a wide population
European Organisation for Research and Treatment of Cancer Questionnaire | At the day of enrollment
  It consists of 30 items and includes three subscales for to assess disease spesific quality of life: global health status, functional status, and symptom control.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Saka, PhD, Study Director — Haliç University
Locations (2):
- Turkey (Türkiye) (2):
  - Halic University, Istanbul
  - Yeditepe Hospital, Istanbul